CLINICAL TRIAL: NCT06506461
Title: St. Jude Autologous Genome Edited Stem Cells For Sickle Cell Disease-1
Brief Title: Gene Editing For Sickle Cell Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAGES1; U01HL163983 (NIH)
Record Dates: First submitted 2024-06-14; First posted 2024-07-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Sickle Cell Disease
Keywords: Plerixafor; Autologous; CD34+ cells; Apheresis; Conditioning; Busulfan; Gene Editing
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — plerixafor; Busulfan

STUDY DESIGN:
Intervention Model Description: Patients with severe sickle cell disease (SCD)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous, genetically modified CD34+ HSPCs Treatment (Experimental): All eligible participants receive intervention as described in the Detailed Description with the following: motixafortide, plerixafor, busulfan, and autologous, gene-modified CD34+ cells
  Interventions: Drug: Plerixafor; Drug: Busulfan; Biological: Gene-modified CD34+ cells; Drug: Motixafortide

INTERVENTIONS:
Drug: Plerixafor — Given Subcutaneous (under the skin)
  Other Names: Mozobil®
Drug: Busulfan — Given Intravenous (IV)
  Other Names: Myleran®; Busulfex
Biological: Gene-modified CD34+ cells — Given Intravenous (IV)
Drug: Motixafortide — Given Subcutaneous (under the skin)
  Other Names: Aphexda

SUMMARY:
This study is being done to test the safety of a new treatment called gene editing in Sickle Cell Disease (SCD) patients and to see if a single dose of this genetically modified cellular product will increase the amount of a certain hemoglobin called fetal hemoglobin (HbF) and help reduce the symptoms of SCD.

Primary Objective

* To assess the safety of autologous infusion of clustered regularly interspaced palindromic repeats (CRISPR)/ CRISPR associated protein (Cas9)-edited CD34+ hematopoietic stem and progenitor cells (HSPCs) in patients with severe SCD.

Secondary Objective

* To assess the efficacy autologous infusion of CRISPR/Cas9 genome-edited CD34+ HSPCs into patients with severe SCD.

DETAILED DESCRIPTION:
Participants will receive a daily subcutaneous (under the skin) dose of motixafortide for up to 3 consecutive days to mobilize their hematopoietic stem and progenitor cells (HSPCs) into peripheral blood. Participants who cannot tolerate motixafortide may receive a daily subcutaneous dose of plerixafor (Mozobil®) as an alternative for 3-5 consecutive days. About 2-4 hours after each dose of plerixafor/motixafortide is given, the collection of HSPCs will start via apheresis. The collected HSPCs will be sent to a lab to genetically modify them using CRISPR/Cas9.

In the lab, the researchers will take the stem cells and purify them. The stem cells will then be mixed with the CRISPR-Cas9 gRNA ribonucleoprotein (RNP) complex to change (edit) the genes in the cells and produce the new gene edited cellular product. This gene edited drug product will be frozen until ready for infusion.

Once the cellular product is ready, participants will be given Busulfan (a chemotherapy medicine) intravenously (IV) for 4 days. The thawed gene product will be given IV about 48 hours after the completion of the last dose of busulfan.

Participants will be followed for 3 years on this study. After the three years, participants will be followed for 12 more years on a long-term follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤24.9 years.
* Patients with SCD (Hb SS, Hb SB0 and Hb SB+ genotype) who have experienced EITHER (a) 2 or more SCD-related vaso-occlusive events (acute pain events, acute chest syndrome, priapism and splenic sequestration) per year in the 2-year period before screening, OR (b) administration of regular red blood cell (RBC) transfusions (≥8 transfusions in the 12 months preceding enrollment) EXCEPT if the RBC transfusions are being administered for primary or secondary stroke prevention and, in the opinion of the treating hematologist, cannot be safely discontinued after infusion of the gene modified drug product.
* Failure, intolerance, or refusal of hydroxyurea therapy.
* Patients must be eligible for autologous stem cell transplant as per investigator's judgment.
* Females of childbearing potential (i.e., those who are post-menarchal with an intact uterus and at least 1 ovary, and those who are less than 1 year postmenopausal) must agree to use acceptable method(s) of contraception from start of mobilization through at least 6 months post-infusion.
* Males must agree to use effective contraception from start of mobilization through at least 6 months post-infusion.
* Patients should be willing to participate in an additional long-term follow-up study after completion of this trial.

Exclusion Criteria:

* Availability of an human leukocyte antigen (HLA)-matched sibling who is willing and able to donate an appropriate graft for hematopoietic cell transplantation (HCT).
* Karnofsky or Lansky performance score < 80.
* Pregnant, as confirmed by positive serum or urine pregnancy test within 14 days before enrollment (if female).
* Breastfeeding.
* Uncontrolled (undergoing appropriate treatment and with progression of clinical symptoms) or clinically significant bacterial, viral, or fungal infections within 1 month before enrollment.
* Patients with confirmed Hepatitis B or Hepatitis C infections.
* Patients with confirmed seropositivity or positive nucleic acid amplification test (NAAT) for human immunodeficiency virus (HIV) or human T-cell lymphotropic virus (HTLV).
* Patients with a history of stroke.
* Serum conjugated (direct) bilirubin > 2× the upper limit of normal for age, or serum alanine transaminase (ALT) > 3× the upper limit of normal for age as per the local laboratory. Participants with hyperbilirubinemia or elevated aspartate aminotransferase (AST) as the result of hyperhemolysis, or with a severe drop in hemoglobin post blood transfusion, are not excluded as long as these values downtrend and return to acceptable limits subsequently.
* Left ventricular shortening fraction < 25% or ejection fraction < 45% by echocardiogram.
* Estimated creatinine clearance less than 60 mL/min/1.73m^2.
* Diffusion capacity of carbon monoxide (DLCO) < 50% (adjusted for hemoglobin) OR baseline oxygen saturation < 85% in patients unable to perform pulmonary function tests.
* Prior HCT or gene therapy.
* Known hepatic cirrhosis, bridging hepatic fibrosis, or active hepatitis. Appropriate ultrasound or magnetic resonance (MR) imaging may be used to define the presence and degree of cirrhosis. Liver biopsy may be performed at the discretion of the attending physician or principal investigator if there are concerns regarding the presence of severe hepatic fibrosis or cirrhosis such that participation in this trial will not be in the patient's best interest.
* Active known malignancy, myelodysplasia, abnormal cytogenetics, or immunodeficiency.
* Patients with history of a significant bleeding disorder.
* Cerebrovascular procedure within 6 months, including pial synangiosis for moyamoya.
* Patients with history of untreated moyamoya disease or presence of moyamoya disease at screening that in the opinion of the investigator puts the subjects at the risk of bleeding.
* Evidence of a pathogenic clonal variant in any candidate gene detected by a standard, licensed next-generation sequencing clinical assay for gene mutations associated hematological malignancies.
* Patients with history of intolerance, contraindication, or known sensitivity to plerixafor or motixafortide or busulfan. Prior anaphylactic reaction with excipients of the proposed product.
* Patients with participation in another clinical study with an investigational drug/product within 30 days of screening or fewer than 5 half-lives of the investigational agent whichever is longer from screening.
* Patients with history of alloimmunization to RBC antigens and for whom the investigator anticipates that there will be insufficient RBC units available for the duration of the study.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of neutrophil engraftment by day +42 after infusion of the CRISPR/Cas9-edited CD34+ HSPCs. | Within 42 days of the cellular product infusion
  Upon completion of the trial, summary statistics will be computed for the time to neutrophil engraftment.
Incidence of platelet engraftment by day +60 after infusion of the CRISPR/Cas9-edited CD34+ HSPCs. | Within 60 days of the cellular product infusion
  Upon completion of the trial, summary statistics will be computed for the time to platelet engraftment.
Sustenance of multi-lineage engraftment and polyclonal hematopoiesis as measured by counts of different clones of myeloid cells, T cells, B cells, and NK cells at 1 year after infusion of the CRISPR/Cas9-edited CD34+ HSPCs. | Within 1 year of the cellular product infusion
  Sustenance of multi-lineage engraftment will be described using descriptive statistics.
Frequency of off-target editing after infusion of the CRISPR/Cas9-edited CD34+ HSPCs. | Within 3 years of the cellular product infusion
  Frequency of off-target editing will be described using descriptive statistics.
Occurrence of secondary graft failure, clonal hematopoiesis, MDS, or AML | Within 3 years of the cellular product infusion
  Occurrence will be described using descriptive statistics.

SECONDARY OUTCOMES:
Estimate the change in the annualized rate of SCD-related vaso-occlusive events (such as pain crises and acute chest syndrome events), starting at 3 months after the infusion of autologous CRISPR/Cas9-edited CD34+ HSPCs. | From 3 months post the cellular product infusion to 3 years post infusion
  We will evaluate the change in the annualized rate of SCD-related vaso-occlusive events starting at 3 months after the infusion of autologous gene-edited CD34+ HSPCs relative to the annualized rate calculated during the 2-year period before study enrollment. The changes will be summarized using descriptive statistics and displayed graphically.
Compare the change from baseline in the total blood hemoglobin concentration. | From time of screening to 3 years post infusion
  The change from baseline (at the time of screening) in the total blood hemoglobin concentration will be calculated at various timepoints as described in the protocol. The changes will be summarized using descriptive statistics and displayed graphically.
Compare the change from baseline in the fraction of red blood cells (RBCs) containing HbF. | From time of screening to 3 years post infusion
  The change from baseline (at the time of screening) in the fraction of RBCs containing HbF by immunostaining will be calculated at various timepoints as described in the protocol. The changes will be summarized using descriptive statistics and displayed graphically.
Change in incidence of packed RBC transfusions. | Within 1 year prior to infusion and within 3 months to 1 year post infusion
  The change from baseline (at the time of screening) in the incidence of packed RBC transfusions will be calculated at various timepoints as described in the protocol. The changes will be summarized using descriptive statistics and displayed graphically.

CONTACTS AND LOCATIONS:
Overall Officials: Akshay Sharma, MBBS, MSc, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — https://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols